CLINICAL TRIAL: NCT01950234
Title: Treatment of Progressive Forms of Multiple Sclerosis With Pulsed ACTH (Acthar Gel)
Brief Title: ACTH in Progressive Forms of MS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funding source discontinued financial support for the study.
Sponsor: University of Minnesota (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110271
Record Dates: First submitted 2013-08-30; First posted 2013-09-25 (Estimated); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Progressive Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACTH (Experimental): ACTH administered subcutaneously as a pulsed regimen of 3 consecutive days per month
  Interventions: Drug: ACTH
- Placebo (Placebo Comparator): Placebo subcutaneous injections administered on 3 consecutive days per month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACTH — Acthar gel
  Other Names: Acthar gel
  Arms: ACTH
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase II, randomized, double-blind, placebo-controlled, multi-center study to evaluate the safety, tolerability, and efficacy of adrenocorticotropic hormone (ACTH, Acthar gel) administered as a pulsed regimen consisting of injections on three consecutive days per month in patients with progressive forms of Multiple Sclerosis (MS). Patients will be randomly assigned to either an ACTH arm or a placebo arm. The main hypotheses are that 1) pulsed ACTH will be safe and well-tolerated, and 2) pulsed ACTH will slow progression of clinical and paraclinical measures of MS progression compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a confirmed diagnosis of MS by McDonald criteria
* Age >/= 18 years
* SPMS, PPMS, or PRMS phenotype, according to Lublin and Reingold criteria
* EDSS 2.0 - 6.0, inclusive
* Able to understand the consent process

Exclusion Criteria:

* Known intolerance of ACTH or corticosteroids
* Diabetes mellitus, defined as pre-existing diagnosis, fasting blood glucose > 125 mg/dl, or glycosylated hemoglobin >/= 6.5%
* Osteoporosis, defined as pre-existing diagnosis or T-score on dual-energy x-ray absorptiometry (DEXA) scan of </= -2.5.
* Current serious medical condition which may interfere with subject's ability to complete the study, or for which pulsed ACTH therapy is contraindicated or might complicate current therapy (e.g., cancer, severe psychiatric illness, chronic infections, autoimmune disorders)
* Treatment with cytotoxic agents (including but not necessarily limited to mitoxantrone, cyclophosphamide, alemtuzumab, or rituximab) within 3 years prior to randomization
* Treatment with non-cytotoxic immunosuppressive agents (including but not necessarily limited to corticosteroids, ACTH, azathioprine, mycophenolate mofetil, methotrexate or natalizumab) within 3 months prior to randomization
* Treatment with FDA-approved first-line MS disease-modifying therapies (B-interferon, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate) will be permitted, as long as treatment has been ongoing and stable for at least 3 months prior to randomization
* Treatment with dalfampridine or compounded 4-aminopyridine (4-AP) will be permitted as long as treatment has been ongoing and stable for at least 3 months prior to randomization
* Stimulant medications for fatigue (such as methylphenidate, modafinil, armodafinil, amantadine or dextroamphetamine) will be permitted, but subjects will be asked to not take these medications on study visit days until all study procedures/assessments are completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam F Carpenter, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Clinical Neuroscience Research Unit, University of Minnesota, Minneapolis, Minnesota
  - Sanford Clinic Neuroscience, Fargo, North Dakota
  - Wheaton Franciscan Healthcare - St Francis Center for Neurological Disorders, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACTH | Placebo
Started | 29 | 30
Completed | 11 | 9
Not Completed | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTH | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.3) | 51.5 (10.2) | 53.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 29 | 58
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Exhibiting a 20% Worsening in T25FW at 36 Months
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 14 | 9
Participants | 3 | 4

2. Secondary Outcome: Safety and Tolerability of ACTH: Menstrual Changes [Female]
Description: Count of participants self reporting at any time throuhgout the study noticing any changes in menstrual cycle or period.
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 12 | 11
Participants | 1 | 1

3. Secondary Outcome: Safety and Tolerability of ACTH: DEXA Scans
Description: The number is a T-score. There is no maximum or minimum value. Mean change in average of 5 DEXA scan values dual-energy x-ray absorptiometry; measures bone mineral density. Higher numbers are better.
  A DEXA T-score has a mean of 0 and standard deviation of 1, meaning that a T-score represents how many standard deviations a person's bone density is away from the average bone density of a healthy young adult, with a score of 0 indicating average bone density. Higher scores are better, indicating better bone density. A T-score of -1 to +1 is considered normal bone density, a score between -1 and -2.5 indicates osteopenia (low bone mass), and a score of -2.5 or lower indicates osteoporosis.
Time Frame: Month 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 14 | 10
units on a scale | -0.41 (0.49) | 0 (0.5)

4. Secondary Outcome: Safety and Tolerability of ACTH: Bruising
Description: Count of participants self reporting at any time throuhgout the study that they bruise more easily
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 7 | 8

5. Secondary Outcome: Safety and Tolerability of ACTH: Swelling Ankles
Description: Count of participants self reporting at any time throuhgout the study that have noticed swelling in their ankles
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 15 | 9

6. Secondary Outcome: Safety and Tolerability of ACTH: Hair Loss
Description: Count of participants self reporting at any time throuhgout the study that have noticed losing more hair
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 7 | 7

7. Secondary Outcome: Safety and Tolerability of ACTH: Acne
Description: Count of participants self reporting at any time throuhgout the study that have noticed in increase in acne
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 2 | 4

8. Secondary Outcome: Safety and Tolerability of ACTH: Insomnia
Description: Count of participants self reporting at any time throuhgout the study that they have been having trouble sleeping
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 12 | 11

9. Secondary Outcome: Safety and Tolerability of ACTH: Mood Change
Description: Count of participants self reporting at any time throuhgout the study that they have noticed changes in mood
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 12 | 11

10. Secondary Outcome: Safety and Tolerability of ACTH: GI Upset
Description: Count of participants self reporting at any time throuhgout the study that they have had upset stomach, indigestion, diarrhea, or bloating
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 5 | 7

11. Secondary Outcome: Safety and Tolerability of ACTH: Fatigue
Description: Count of participants self reporting at any time throuhgout the study that noticed feeling tired or worn out
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 16 | 14

12. Secondary Outcome: Safety and Tolerability of ACTH: Unpleasant Taste
Description: Count of participants self reporting at any time throuhgout the study noticing a metallic taste in their mouth
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 4 | 3

13. Secondary Outcome: Safety and Tolerability of ACTH: Blurred Vision
Description: Count of participants self reporting at any time throuhgout the study noticing any blurred vision
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 4 | 7

14. Secondary Outcome: Safety and Tolerability of ACTH: Moon Facies
Description: New physician assessed moon facies over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

15. Secondary Outcome: Safety and Tolerability of ACTH: Skin Thinning
Description: New physician assessed skin thinning over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 3 | 3

16. Secondary Outcome: Safety and Tolerability of ACTH: Hirsuitism
Description: New physician assessed hirsuitism over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 1 | 1

17. Secondary Outcome: Safety and Tolerability of ACTH: Bruising
Description: New physician assessed bruising over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 4 | 4

18. Secondary Outcome: Safety and Tolerability of ACTH: Ankle Swelling
Description: New physician assessed ankle swelling over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 7 | 5

19. Secondary Outcome: Safety and Tolerability of ACTH: Hair Loss
Description: Any new physician assessed hair loss over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 4 | 3

20. Secondary Outcome: Safety and Tolerability of ACTH: Cataracts
Description: New physician assessed cataracts over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 2 | 1

21. Secondary Outcome: Safety and Tolerability of ACTH: Myopathy
Description: New physician assessed myopathy over study duration
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

22. Secondary Outcome: Safety and Tolerability of ACTH: Change in Hemoglobin A1c
Description: Change in hemoglobin A1c
Time Frame: Month 36
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | ACTH | Placebo
Number analyzed (Participants) | 14 | 10
percent | 0.14 (0.36) | 0.05 (0.32)

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | ACTH | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 8/29 | 7/30
Other Adverse Events (participants affected / at risk) | 29/29 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTH (N=29) | Placebo (N=30)
Gastrointestinal (Gastrointestinal disorders) | 4 (6) | 2 (3)
infection (General disorders) | 2 (2) | 3 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTH (N=29) | Placebo (N=30)
Alopecia (General disorders) | 4 (4) | 6 (7)
Bladder function (Renal and urinary disorders) | 5 (5) | 2 (2)
Bruising (General disorders) | 7 (7) | 11 (11)
cardiovascular (Cardiac disorders) | 14 (17) | 8 (10)
dermatologic (General disorders) | 7 (10) | 10 (12)
Dysgeusia (General disorders) | 4 (4) | 2 (2)
Edema (General disorders) | 14 (24) | 9 (10)
Fatigue (General disorders) | 12 (12) | 12 (12)
Gastrointestinal (Gastrointestinal disorders) | 9 (26) | 13 (15)
genitourinary (General disorders) | 0 (0) | 2 (3)
Infection (General disorders) | 9 (25) | 13 (22)
Injection site reaction (General disorders) | 3 (12) | 6 (6)
Metabolic (General disorders) | 3 (3) | 0 (0)
Metabolic/endocrine (General disorders) | 6 (8) | 5 (5)
Mood (General disorders) | 11 (14) | 11 (12)
Musculoskeletal (General disorders) | 22 (83) | 16 (46)
Neoplasm (General disorders) | 4 (6) | 0 (0)
Neurologic (Nervous system disorders) | 15 (38) | 9 (17)
other (General disorders) | 9 (14) | 2 (2)
renal (Renal and urinary disorders) | 0 (0) | 1 (3)
respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
sleep (General disorders) | 14 (19) | 9 (9)
visual (General disorders) | 13 (16) | 8 (11)
weight gain (General disorders) | 8 (10) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT01950234/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT01950234/ICF_001.pdf